CLINICAL TRIAL: NCT06159270
Title: Collection of Prospective Biological Samples for Biological Analysis in Current Clinical Practice
Brief Title: Infectious Prospective Collection for Biological Analysis
Acronym: Infectieux1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CerbaXpert (Other)
Responsible Party: Sponsor
Other Study IDs: Infectieux 1
Record Dates: First submitted 2023-11-17; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Infectious Disease
MeSH Terms: conditions — Communicable Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of patients presenting infectious diseases
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Venuous blood sampling

SUMMARY:
The increase in activity within medical biology laboratories linked to the arrival of new markers (in cardiology, oncology, infectious diseases, etc.) and the acceleration of technical progress have created a prominent place for automated systems and their reagent kits within these establishments.

It is in this context that CerbaXpert took the initiative to set up this research project for the collection of prospective biological samples and their analysis. It transcribes both a process of continuous improvement but also scientific development, making it possible to provide new and/or complementary data in order to improve the operation of automated systems and their reagents within medical biology laboratories. These data obtained in current practice via this study will also be compared with the technical information provided by the manufacturers of the reagents and their automatic devices.

DETAILED DESCRIPTION:
This research protocol is a prospective multicenter collection of biological samples for evaluation of reagents and automated systems on the following parameters: HAV, B, C, D and E, HIV, HBV, EBV, CMV, VZV, HPV, HSV, polyomavirus family, Chlamydia Trachomatis, Neisseria gonorrhoeae, Mycoplasma genitalium, Trichomonas vaginalis, Treponema pallidum, Zika virus, dengue fever, chikungunya virus, influenza virus, Mycobacterium tuberculosis bacteria, parasite responsible for toxoplasmosis, malaria, rubella virus, Lyme borreliosis Sars-CoV-2 virus responsible for Covid-19 disease, bacteria responsible for leptospirosis and salmonellosis, the pathogens responsible for sepsis (viruses, bacteria or fungus) and finally the Poxiviridae family. This research is categorized as Research Involving Human Person level 3 (RIPH 3), that is to say non-interventional, carried out in current medical practice. Recruitment will include a maximum of 22870 samples belonging to the following groups: population general (ambulatory patients, hospitalized patients, pregnant women, dialysis patients) and known population carrying the desired infectious agent.

This protocol does not include special procedure for allocation or differential treatment for the subjects included: there is neither randomization or treatment assigned to people participating in the study.

The subjects recruited will be within several survey sites spread across the national territory: the Cerballiance medical biology laboratories, belonging to the Cerba HealthCare group. Some clinical sites can be managed via a centralized collection site, where a person is designated as principal investigator after qualification by the promoter and authorization from the Committee of Protection of People.

Information relating to age, sex, date and place of sampling, sample population of each subject (general patients, hospitalized patients, pregnant women, dialysis patients or patients known positive for one of the infectious agents targeted by this research protocol) will be also varied. Relevant medical data may also be compiled:

1. the genotype of HAV, B, C, D and E, HIV, HBV (if available);
2. the stage of the disease (acute, chronic, cured);
3. concomitant treatments linked to the pathology (if available) or which may interfere with the planned analysis.
4. data relating to the participant's lifestyle.
5. date of onset of symptoms, date of PCR test if applicable, vaccination status, date of vaccination, name of vaccine, number of injections, batch number of vaccine.

ELIGIBILITY:
Inclusion Criteria:

* All-comers clinical subjects (ambulatory)
* Hospitalized patients
* Pregnant women (all comers)
* Subjects on dialysis
* Known subjects positive for targeted pathogens

Exclusion Criteria:

* Subject having already participated in this protocol within 15 days previous ones.
* Subject having received medication or treatment experimental or investigational during the last four weeks before collection
* Person subject to a judicial safeguard measure
* Person not affiliated to the Social Security system and not not having social security coverage
* Person not meeting the inclusion criteria

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Man or woman, aged 18 to 88, coming for an analysis biological as part of routine care, for prevention, screening or the monitoring of at least one of the pathogens targeted or benefiting of a teleconsultation and accepting additional samples carried out by a healthcare professional and, where applicable, capable of allow a maximum of 21 ml of whole blood or two swabs additional and able to give consent
Sampling Method: Non-Probability Sample
Enrollment: 22870 (Estimated)
Dates: Start 2019-05-18 (Actual); Primary Completion 2025-05-18 (Estimated); Study Completion 2025-05-18 (Estimated)

PRIMARY OUTCOMES:
Evaluation of clinical and analytical performance of In vitro diagnostic tests used in routine care for infectious diseases by using ROC curve | 24 months
  * Venipuncture sampling
  * Blood sampling by capillary action
  * Swab sampling
  * Salivary samples
  * Urine sampling
  * Dried Blood Spot (DBS) sampling

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Pernicni, Dr, Study Director — Cerba Xpert
Locations (1):
- Cerba Xpert, Saint-Ouen-l'Aumône, France

IPD SHARING:
Plan to Share IPD: No